CLINICAL TRIAL: NCT04214353
Title: Effect of Androgen Deprivation Therapy on Uptake of PSMA Ligand in Patients With Salivary Duct Carcinoma: an Explorative Study.
Brief Title: PSMA-PET Imaging Before and After ADT in Advanced SDC Patients
Acronym: ADT-SCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MOHN19
Record Dates: First submitted 2019-12-13; First posted 2020-01-02 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Salivary Gland Cancer; Salivary Duct Carcinoma
Keywords: Positron-Emission Tomography; 68Ga-PSMA-PET/CT; 18FDG-PET/CT; Androgen deprivation therapy
MeSH Terms: conditions — Salivary Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Salivary duct carcinoma patients with R/M disease, who will start androgen deprivation therapy as standard of care will receive PET/CT scans before and after ADT.
  Interventions: Diagnostic Test: 68Ga-PSMA-PET/CT; Diagnostic Test: 18FDG-PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-PET/CT — All participants in the study will be injected with 2.0 MBq/kg 68Ga-PSMA for PET/CT imaging, both pre- and post ADT.
Diagnostic Test: 18FDG-PET/CT — All participants in the study will be injected with 2.1 MBq/kg 18FDG for PET/CT imaging, both pre- and post ADT.

SUMMARY:
Explorative study, which evaluates the effect of androgen deprivation therapy (ADT) on the PSMA ligand uptake on 68Ga-PSMA-PET/CT in salivary duct carcinoma patients.

DETAILED DESCRIPTION:
Rationale: Prostate specific membrane antigen (PSMA) is a transmembrane protein, which is expressed on prostate cancers cells and other malignancies. Recently, several ligands have been developed that target PSMA. Linked to Gallium-68, this enables diagnostic 68Ga-PSMA-PET/CT scans. Linked to Lutetium-177 enables therapeutic 177Lu-PSMA Radioligand therapy. Most research on the diagnostic and therapeutic possibilities of PSMA has been conducted in patients with advanced prostate cancer.

This research group investigates whether these findings also apply to salivary gland cancer (SGC), a rare cancer. Previously the investigators conducted a phase II 68Ga-PSMA imaging study (NCT03319641), to evaluate PSMA ligand uptake in locally advanced, recurrent and metastatic ACC and SDC (two subtypes of SGC). A relevant PSMA-ligand uptake was observed in 93% of ACC patients and 40% of SDC patients. However, since 60% of SDC patients showed low ligand uptake, these patients are not suitable for PSMA radioligand therapy. For advanced SDC, androgen deprivation therapy is often given as first-line treatment, because the majority of SDCs are androgen receptor positive. In prostate cancer, androgen deprivation therapy (ADT) can increase PSMA-ligand uptake. Therefore the aim is to investigate if ADT can increase the uptake of 68Ga-PSMA in patients with R/M SDC, as has previously been demonstrated in prostate cancer.

Objective: The primary objective is to investigate if ADT can increase the uptake of 68Ga-PSMA in patients with R/M SDC.

Study design: Interventional clinical trial, an explorative study. Study population: Patients with locally advanced, recurrent or metastatic (R/M) SDC AR+ and who will start ADT as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to provide written informed consent.
* Patients must be ≥ 18 years of age.
* Patients must have histological, pathological, and/or cytological confirmation of salivary duct carcinoma, androgen receptor positive.
* Only patients with locally advanced, recurrent or metastatic salivary duct carcinoma can participate.
* Patients must have at least one lesion with a diameter of ≥ 1.5 cm.
* Patients whom intend to start androgen deprivation therapy, after this has been recommended by the treating physician as standard treatment.

Exclusion Criteria:

* Contra-indication for PET imaging (pregnancy, breast feeding severe claustrophobia)
* Impaired renal function: MDRD <30 ml/min/1,73 m2
* Impaired liver function: AST and ALT ALT ≥ 2.5 x ULN (≥5 x ULN for patients with liver metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a change in PSMA ligand uptake after ADT | Up to 4 weeks
  The percentage of patients with an androgen deprivation therapy (ADT) induced change in PSMA ligand uptake on 68Ga-PSMA-PET/CT.
  pre-scan: baseline (before ADT), post-scan: 3 weeks after start ADT (± 1 week).

SECONDARY OUTCOMES:
Change in 68Ga-PSMA uptake of tumor lesions | Up to 4 weeks
  Comparison of SUV (standardized uptake value) in 68Ga-PSMA PET/CT between lesions before and 3 weeks after the initiation of ADT (± 1 week).
Change in 18FDG uptake of tumor lesions | Up to 4 weeks
  Comparison of SUV (standardized uptake value) in 18FDG-PET/CT between lesions before and 3 weeks after the initiation of ADT (± 1 week).
Lesions detected by 68Ga-PSMA-PET/CT pre- and post ADT | Up to 4 weeks
  The number of lesions detected on 68Ga-PSMA-PET/CT imaging will be measured, both before and after ADT.
FDG and PSMA uptake patterns of SDC disease | Up to 4 weeks
  FDG and PSMA uptake patterns of SDC disease on 68Ga-PSMA-PET/CT and 18FDG-PET/CT will be measured, e.g. to explore if most lesions show both FDG and PSMA uptake, or if the lesions show a more heterogenous uptake.
Diagnostic added value 68Ga-PSMA-PET/CT and 18FDG-PET/CT. | Up to 4 weeks
  The number of lesions detected by each imaging modality (diagnostic CT, 68Ga-PSMA-PET/CT and 18FDG-PET/CT) will be measured.
Correlation PSMA expression and PSMA ligand uptake | Up to 6 months
  The tumor uptake (SUV) will be correlated to the degree of immunohistochemical PSMA expression on the most recent tumormaterial.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Ruitenbeek NJ, Uijen MJM, Driessen CML, van Rijk MC, Peters SMB, Prive BM, Verhaegh GW, van Engen-van Grunsven ACH, Gotthardt M, Nagarajah J, van Herpen CML. The effect of androgen blockade on [68Ga]Ga-PSMA-11 and [18F]FDG PET uptake in patients with recurrent or metastatic salivary duct carcinoma: a prospective imaging study. EJNMMI Res. 2025 Jul 15;15(1):86. doi: 10.1186/s13550-025-01275-x. PMID 40663212